CLINICAL TRIAL: NCT03931109
Title: Circulating microRNA Signatures in Primary Hyperparathyroidism
Brief Title: Circulating miRNA in Primary Hyperparathyroidism
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 829615
Record Dates: First submitted 2019-04-15; First posted 2019-04-30 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-04

CONDITIONS: Primary Hyperparathyroidism; Osteoporosis, Postmenopausal
Keywords: Osteoporosis; primary hyperparathyroidism; miRNA; Bone remodeling; parathyroidectomy; Osteopenia; postmenopausal
MeSH Terms: conditions — Hyperparathyroidism, Primary; Osteoporosis, Postmenopausal; Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PHPT w/ Osteoporosis: Primary hyperparathyroidism patients with osteoporosis undergoing parathyroidectomy
- PHPT w/o Osteoporosis: Primary hyperparathyroidism patients without osteoporosis undergoing parathyroidectomy
- Thyroid w/ Osteoporosis: Thyroid disease patients with osteoporosis undergoing thyroidectomy

SUMMARY:
The goal of this study is to: 1. Analyze the expression levels of circulating (serum) miRNAs in primary hyperparathyroidism patients with and without osteoporosis, and patients with osteoporosis undergoing thyroidectomy, and to correlate with clinical markers of bone remodeling including biochemical and radiologic studies. 2. To evaluate serum miRNA levels after treatment with parathyroidectomy.

DETAILED DESCRIPTION:
Osteoporosis and osteopenia are chronic diseases disproportionately affecting the elderly. In the United States, the prevalence of osteoporosis is projected to increase from 10 million in 2005 to 14 million in 2025, due to population aging. Similarly, the economic cost of osteoporotic fractures is projected to increase to $25 billion by 2025. Primary hyperparathyroidism (PHPT) is one of the few reversible causes of osteoporosis and fragility fractures. PHPT is the third most common endocrine disorder, with an incidence of 27-30 per 100,000 person-years, and increasing with age; half of all patients with PHPT are post-menopausal women, a population at high risk for osteoporosis at baseline. All forms of PHPT are characterized by loss of the normal negative feedback relationship between serum calcium and parathyroid hormone (PTH) secretion, leading to hypercalcemia and hyperparathyroidism. Classic PHPT is characterized by skeletal, renal, gastrointestinal and neuropsychiatric manifestations. Skeletal manifestations of classic PHPT are mediated by osteoblast inhibition and osteoclast stimulation, leading to increased bone remodeling. The catabolic effects of chronic PTH excess may present as osteitis fibrosa cystica, brown tumors, pathologic fractures, bone pain, osteoporosis or osteopenia. Although frank osteitis fibrosa cystica is an increasingly rare presentation of PHPT in the United States, affecting 2% of patients, osteoporosis is reported in 39-63% of patients, with preferential loss of bone density in cortical sites. Fragility fractures are significantly associated with PHPT, particularly in postmenopausal women. Both decreases in bone mineral density (BMD) and fragility fractures are considered indications for parathyroidectomy in patients with asymptomatic PHPT. Parathyroidectomy has been demonstrated to improve BMD in prospective studies of PHPT patients with osteoporosis; some studies suggest that more benefit may be seen in pre-menopausal women. Current research in bone remodeling has identified microRNAs (miRNAs), novel biomarkers with both diagnostic and therapeutic potential. miRNAs are short, single stranded, non-coding RNAs which regulate posttranscriptional expression of mRNA. miRNAs have been extensively implicated in bone remodeling and homeostasis. Circulating miRNAs have been shown to correlate with fragility fractures, and are conserved across subpopulations of osteoporotic patients. miRNA panels have been suggested to have the potential to assist in diagnosis, prognosis, and are promising targets for directed therapy. Although miRNAs have been investigated in conjunction with pre-menopausal, postmenopausal, idiopathic and diabetic osteoporosis, no research to date has explored the miRNA profile of PHPT patients with osteoporosis. Similarly, although in vitro experiments have demonstrated miRNA response to bisphosphonates, no clear correlation has been established between therapeutic interventions and miRNA levels in vivo. The goal of this study is therefore two-fold; first, to analyze the expression levels of circulating miRNAs in PHPT patients with and without osteoporosis; and second, to evaluate miRNA levels after treatment with parathyroidectomy.

This is a prospective, non-randomized pilot study. Post-menopausal female subjects with and without osteoporosis, undergoing neck surgery or non-operative management will be recruited. Informed consent will be obtained. Venipuncture will be performed and serum and plasma isolated from study subjects. Analysis of serum miRNA and biochemical and clinical markers of bone remodeling will be performed. Clinical care will proceed as planned. Subjects undergoing surgery will be reassessed one year after operative intervention for miRNA and clinical and biochemical markers.

ELIGIBILITY:
Inclusion Criteria:

* post menopausal
* has had DXA scan
* has 24 hr Urine Calcium
* Elevated serum calcium
* Vitamin D above 20 ng/ml
* capable of giving informed consent
* female
* indication for biochemical primary hyperparathyroidism or an indication for partial or total thyroidectomy

Exclusion Criteria:

* history of ESRD on dialysis or renal osteodystrophy
* prior parathyroidectomy
* hyper or hypothyroid by TSH
* currently taking steroids or has been on steroids for more than 7 days in the last two years
* estrogen therapy within the last two years
* bisphosphonate therapy within the last two years
* diagnosis of Cushing's disease or Cushing's syndrome
* taking biotin within 24 hours of blood draw

Ages: 50 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: post-menopausal women diagnosed with primary hyperparathyroidism.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
circulating microRNAs in primary hyperparathyroidism patients | 2019-2021
  Serum miRNA levels
serum miRNA after parathyroidectomy | 2019-2021
  clinical markers of bone remodeling, including serum levels of bone-specific alkaline phosphatase, osteocalcin, P1NP, CTX, calcium, phosphate, Vitamin D metabolites, and PTH; urine calcium; and DXA scan

CONTACTS AND LOCATIONS:
Overall Officials: Heather Wachtel, MD, Principal Investigator — University of Pennsylvania Health System
Locations (1):
- Perelman Center for Advanced Medicine/ Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Burge R, Dawson-Hughes B, Solomon DH, Wong JB, King A, Tosteson A. Incidence and economic burden of osteoporosis-related fractures in the United States, 2005-2025. J Bone Miner Res. 2007 Mar;22(3):465-75. doi: 10.1359/jbmr.061113. PMID 17144789
- [Background] Fraser WD. Hyperparathyroidism. Lancet. 2009 Jul 11;374(9684):145-58. doi: 10.1016/S0140-6736(09)60507-9. PMID 19595349
- [Background] Lewiecki EM, Miller PD. Skeletal effects of primary hyperparathyroidism: bone mineral density and fracture risk. J Clin Densitom. 2013 Jan-Mar;16(1):28-32. doi: 10.1016/j.jocd.2012.11.013. PMID 23374738
- [Background] Walker MD, Silverberg SJ. Primary hyperparathyroidism. Nat Rev Endocrinol. 2018 Feb;14(2):115-125. doi: 10.1038/nrendo.2017.104. Epub 2017 Sep 8. PMID 28885621
- [Background] De Geronimo S, Romagnoli E, Diacinti D, D'Erasmo E, Minisola S. The risk of fractures in postmenopausal women with primary hyperparathyroidism. Eur J Endocrinol. 2006 Sep;155(3):415-20. doi: 10.1530/eje.1.02225. PMID 16914595
- [Background] Vignali E, Viccica G, Diacinti D, Cetani F, Cianferotti L, Ambrogini E, Banti C, Del Fiacco R, Bilezikian JP, Pinchera A, Marcocci C. Morphometric vertebral fractures in postmenopausal women with primary hyperparathyroidism. J Clin Endocrinol Metab. 2009 Jul;94(7):2306-12. doi: 10.1210/jc.2008-2006. Epub 2009 Apr 28. PMID 19401378
- [Background] Bilezikian JP, Brandi ML, Eastell R, Silverberg SJ, Udelsman R, Marcocci C, Potts JT Jr. Guidelines for the management of asymptomatic primary hyperparathyroidism: summary statement from the Fourth International Workshop. J Clin Endocrinol Metab. 2014 Oct;99(10):3561-9. doi: 10.1210/jc.2014-1413. Epub 2014 Aug 27. PMID 25162665
- [Background] Lundstam K, Heck A, Godang K, Mollerup C, Baranowski M, Pernow Y, Aas T, Hessman O, Rosen T, Nordenstrom J, Jansson S, Hellstrom M, Bollerslev J; SIPH Study Group. Effect of Surgery Versus Observation: Skeletal 5-Year Outcomes in a Randomized Trial of Patients With Primary HPT (the SIPH Study). J Bone Miner Res. 2017 Sep;32(9):1907-1914. doi: 10.1002/jbmr.3177. Epub 2017 Jul 7. PMID 28543873
- [Background] Lumachi F, Camozzi V, Ermani M, DE Lotto F, Luisetto G. Bone mineral density improvement after successful parathyroidectomy in pre- and postmenopausal women with primary hyperparathyroidism: a prospective study. Ann N Y Acad Sci. 2007 Nov;1117:357-61. doi: 10.1196/annals.1402.012. Epub 2007 Jul 23. PMID 17646261
- [Background] Kim KM, Lim SK. Role of miRNAs in bone and their potential as therapeutic targets. Curr Opin Pharmacol. 2014 Jun;16:133-41. doi: 10.1016/j.coph.2014.05.001. Epub 2014 Jun 5. PMID 24907412
- [Background] Garnero P. New developments in biological markers of bone metabolism in osteoporosis. Bone. 2014 Sep;66:46-55. doi: 10.1016/j.bone.2014.05.016. Epub 2014 Jun 5. PMID 24909537
- [Background] Jing D, Hao J, Shen Y, Tang G, Li ML, Huang SH, Zhao ZH. The role of microRNAs in bone remodeling. Int J Oral Sci. 2015 Sep 14;7(3):131-43. doi: 10.1038/ijos.2015.22. PMID 26208037
- [Background] Heilmeier U, Hackl M, Skalicky S, Weilner S, Schroeder F, Vierlinger K, Patsch JM, Baum T, Oberbauer E, Lobach I, Burghardt AJ, Schwartz AV, Grillari J, Link TM. Serum miRNA Signatures Are Indicative of Skeletal Fractures in Postmenopausal Women With and Without Type 2 Diabetes and Influence Osteogenic and Adipogenic Differentiation of Adipose Tissue-Derived Mesenchymal Stem Cells In Vitro. J Bone Miner Res. 2016 Dec;31(12):2173-2192. doi: 10.1002/jbmr.2897. Epub 2016 Sep 26. PMID 27345526
- [Background] Kocijan R, Muschitz C, Geiger E, Skalicky S, Baierl A, Dormann R, Plachel F, Feichtinger X, Heimel P, Fahrleitner-Pammer A, Grillari J, Redl H, Resch H, Hackl M. Circulating microRNA Signatures in Patients With Idiopathic and Postmenopausal Osteoporosis and Fragility Fractures. J Clin Endocrinol Metab. 2016 Nov;101(11):4125-4134. doi: 10.1210/jc.2016-2365. Epub 2016 Aug 23. PMID 27552543
- [Background] Weilner S, Skalicky S, Salzer B, Keider V, Wagner M, Hildner F, Gabriel C, Dovjak P, Pietschmann P, Grillari-Voglauer R, Grillari J, Hackl M. Differentially circulating miRNAs after recent osteoporotic fractures can influence osteogenic differentiation. Bone. 2015 Oct;79:43-51. doi: 10.1016/j.bone.2015.05.027. Epub 2015 May 28. PMID 26026730
- [Background] Hackl M, Heilmeier U, Weilner S, Grillari J. Circulating microRNAs as novel biomarkers for bone diseases - Complex signatures for multifactorial diseases? Mol Cell Endocrinol. 2016 Sep 5;432:83-95. doi: 10.1016/j.mce.2015.10.015. Epub 2015 Oct 23. PMID 26525415
- [Background] Zhou Q, Zhao ZN, Cheng JT, Zhang B, Xu J, Huang F, Zhao RN, Chen YJ. Ibandronate promotes osteogenic differentiation of periodontal ligament stem cells by regulating the expression of microRNAs. Biochem Biophys Res Commun. 2011 Jan 7;404(1):127-32. doi: 10.1016/j.bbrc.2010.11.079. Epub 2010 Nov 23. PMID 21108928

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT03931109/Prot_SAP_001.pdf
  • Informed Consent Form (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT03931109/ICF_000.pdf